CLINICAL TRIAL: NCT05368961
Title: Comparison of Midazolam (Versed) and Distraction on Anxiety, Emergence Delirium, Sedation/Agitation, and Vomiting in Pre-operative Patients Ages 3 to 5.
Brief Title: Comparison of Usual Care and Distraction (Tablet) in Children 3-5 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michelle Levay, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-511
Record Dates: First submitted 2022-04-28; First posted 2022-05-10 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Intervention Model Description: Group 1: usual care Group 2: distraction
Masking Description: Not a blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Usual care (midazolam) is administered pre-operatively
  Interventions: Other: Usual care
- Distraction (Experimental): Distraction (interactive tablet) is given to children pre-operatively
  Interventions: Behavioral: Distraction

INTERVENTIONS:
Behavioral: Distraction — Distraction (interactive tablet)
  Arms: Distraction
Other: Usual care — Anxiolytic ordered by anesthesiologist is usual care
  Other Names: Anxiolytic per anesthesia
  Arms: Usual care

SUMMARY:
Randomized control trial comparing usual care and distraction (tablet) on anxiety, emergence delirium, sedation/agitation, and vomiting in children 3-5 years old

DETAILED DESCRIPTION:
Two group RCT comparing usual care (midazolam) and distraction (tablet) on preoperative anxiety, emergence delirium, sedation/agitation, and vomiting in preschool children 3-5 years old.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 year old children
* Scheduled for elective surgery
* American Society of Anesthesiologists physical status classification system: I - II

Exclusion Criteria:

* Children younger than 3 or older than 6
* Allergy to midazolam
* Cognitive or developmental delays
* American Society of Anesthesiologists physical status classification system: III - VI
* Anesthesia provider determines child is not eligible
* Children that are transferred to ICU after surgery

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Albert, PhD, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seiden SC, McMullan S, Sequera-Ramos L, De Oliveira GS Jr, Roth A, Rosenblatt A, Jesdale BM, Suresh S. Tablet-based Interactive Distraction (TBID) vs oral midazolam to minimize perioperative anxiety in pediatric patients: a noninferiority randomized trial. Paediatr Anaesth. 2014 Dec;24(12):1217-23. doi: 10.1111/pan.12475. Epub 2014 Jul 17. PMID 25040433
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children ages 3-5 years were recruited from the pre-operative area at a single surgery site between April 2017 to March 2019.
Period: Overall Study
Arm/Group | Usual Care | Distraction
Started | 74 | 63
Completed | 47 | 52
Not Completed | 27 | 11

BASELINE CHARACTERISTICS:
Population: Data was not reported on participants lost to attrition
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Distraction | Total
Number analyzed (Participants) | 47 | 52 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47 | 52 | 99
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Customized [Count of Participants; unit: Participants]
  3 years old | 24 | 22 | 46
  4 years old | 16 | 15 | 31
  5 years old | 7 | 15 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 24 | 39
  Male | 32 | 28 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 39 | 45 | 84
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 2 | 6
Type of surgery [Count of Participants; unit: Participants]
  Ear Nose Throat | 20 | 30 | 50
  Ophthalmology | 13 | 18 | 31
  Urology | 10 | 2 | 12
  General Surgery | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: mYPAS Anxiety Score, Patients With Scores of 30 or More Indicated "Anxiety"
Description: Pre-operative anxiety measured by the modified Yale Preoperative Anxiety Scale (mYPAS); scores range 23-100 with higher scores indicating greater levels of anxiety.
  A categorical variable was created using a cut-off score of 30 or more to indicate "anxiety" and scores of less than 30 indicated "no anxiety".
Time Frame: Pre-induction of mask anesthesia in the operating room
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Distraction
Number analyzed (Participants) | 47 | 52
Participants | 20 | 22
Statistical Analysis 1: Comparison: Usual Care vs Distraction; Test type: Other — Null hypothesis; there is no difference in anxiety scores between usual care and distraction; p = 0.44, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Sedation/Agitation
Description: Sedation/agitation was assessed using the Richmond Agitation Sedation Scale (RASS)
  The RASS scale is a 10-item observational tool. Scores on RASS range from negative 5 (unarousable) to positive 4 (combative/violent). For this study, we categorized the RASS scores as agitated, calm, or sedated. Scores of 2 or higher indicated "agitation", scores of +1 to -1 were "calm", and scores of -2 or lower indicated "sedation".
Time Frame: Pre-induction of mask anesthesia in the operating room
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Distraction
Number analyzed (Participants) | 47 | 52
Participants
  Sedated | 1 | 0
  Calm | 42 | 45
  Agitated | 4 | 7

3. Secondary Outcome: Number of Participants Experiencing Emergence Delirium
Description: Postoperatively pediatric patients were assessed for emergence delirium using the Pediatric Anesthesia Emergence Delirium (PAED) tool.
  The scale uses a 5-point Likert scale with total scores ranging from 0 - 20. This study used a score of 12-20 to indicate the presence of "emergence delirium."
Time Frame: After surgery when patient woke up in the post anesthesia care unit (recovery room)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Distraction
Number analyzed (Participants) | 47 | 52
Participants | 7 | 8

4. Secondary Outcome: Sedation/Agitation
Description: as for outcome 2
Time Frame: After surgery at the time of admission to post anesthesia care unit (recovery room)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Distraction
Number analyzed (Participants) | 47 | 52
Participants
  Sedated | 45 | 48
  Calm | 0 | 3
  Agitated | 2 | 1

5. Secondary Outcome: Length of Stay (Minutes)
Description: Length of stay (total minutes) = time patient admitted to post anesthesia care unit (recovery room) until discharged from post anesthesia care unit.
Time Frame: Post operative until discharged from post anesthesia care unit (recovery room)
Measure: Mean (Inter-Quartile Range); unit: Minutes
Arm/Group | Usual Care | Distraction
Number analyzed (Participants) | 47 | 52
Minutes | 88.0 [78.0 to 101.0] | 75.5 [59.5 to 98.0]

6. Secondary Outcome: The Number of Patients Experiencing Postoperative Vomiting
Description: The number of participants that vomited in the post-anesthesia care unit (from the time they were admitted until they were discharged).
Time Frame: After surgery in the post anesthesia care unit from admission to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Distraction
Number analyzed (Participants) | 47 | 52
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Time in study = time they received the intervention (control or experimental) until discharged from post anesthesia care unit. Each participant was in the study from 2-6 hours. Operating room times varied by surgical procedure.
Description: Not applicable, no adverse events reported.
Arm/Group | Usual Care | Distraction
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/52
Other Adverse Events (participants affected / at risk) | 0/47 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT05368961/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT05368961/SAP_001.pdf